CLINICAL TRIAL: NCT05597163
Title: A Multicenter, Double-blind, Randomized, Controlled Clinical Study of the Efficacy and Safety of Low-concentration Atropine for Myopia Control in Chinese Children and Adolescents
Brief Title: Efficacy and Safety of Low-concentration Atropine for Myopia Control in Chinese Children and Adolescents
Acronym: LAMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Peking University People's Hospital (Other); Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kjb-atp-v1.1-20220825
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-10

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.01% atropine (Experimental): 0.01% atropine eye drop
  Interventions: Drug: low concentration atropine (0.01%)
- 0.025% atropine (Experimental): 0.025% atropine eye drop
  Interventions: Drug: low concentration atropine (0.025%)
- 0.05% atropine (Experimental): 0.05% atropine eye drop
  Interventions: Drug: low concentration atropine (0.05%)
- cross-over (Other): first year: placebo second year: 0.05% atropine eye drop
  Interventions: Drug: low concentration atropine (0.05%); Drug: Placebo

INTERVENTIONS:
Drug: low concentration atropine (0.01%) — 0.01% atropine eye drop
  Arms: 0.01% atropine
Drug: low concentration atropine (0.025%) — 0.025% atropine eye drop
  Arms: 0.025% atropine
Drug: low concentration atropine (0.05%) — 0.05% atropine eye drop
  Arms: 0.05% atropine; cross-over
Drug: Placebo — Placebo eye drop
  Arms: cross-over

SUMMARY:
To investigate the efficacy and safety of three low-concentration atropine sulfate eye drops (0.01%, 0.025% and 0.05%) in controlling the progression of myopia in Chinese children and adolescents through a two-year clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the screening stage is 3-15 years, both sexes;
2. One eye met the diagnosis of myopic refractive error, the spherical equivalent was between -0.50D and -8.00D, the astigmatism was ≥-3.00D, and the best corrected far vision was at least 0.8;
3. Have normal thinking and language communication ability, and can actively cooperate with treatment and follow-up as required;
4. Informed consent from the guardian and the child.

Exclusion Criteria:

1. strabismus, amblyopia or other ocular abnormalities;
2. The presence of systemic disease abnormalities;
3. have taken myopia control treatment in the past month;
4. Allergic to low concentration atropine or sulfuric acid drugs.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 588 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of SE changes over -0.75D | 2 years

SECONDARY OUTCOMES:
AL change | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zou, Study Director — Shanghai Eye Disease Prevention and Treatment Center